CLINICAL TRIAL: NCT06604702
Title: Fat Injection for Treatment of Rectocele a Novel Technique for Treatment of Tectocele
Brief Title: Fat Injection for Rectocele Treatment: A Novel Approach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eslam Mohamed Hagagy Mohamed, Resident of the General Surgery, Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-260-2022
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rectocele; Pelvic Organ Prolapse; Obstructive Defecation Syndrome
Keywords: Rectocele; Pelvic Floor Dysfunction; Fat Grafting; Autologous Fat Injection; Obstructive Defecation; Pelvic Organ Prolapse; Vaginal Bulge
MeSH Terms: conditions — Rectocele; Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Single-arm prospective interventional trial where all participants undergo submucosal fat injections for the treatment of rectocele.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fat Injection for Rectocele (Experimental): Participants in this arm will undergo autologous fat injection as a novel treatment for rectocele. Fat grafts will be harvested from the patient's abdomen, processed to purify the fat, and injected into the submucosal layer of the rectocele through the posterior vaginal wall. This procedure aims to reduce the size of the rectocele, alleviate symptoms like vaginal bulge and obstructive defecation, and prevent recurrence.
  Interventions: Procedure: Autologous Fat Injection for Rectocele

INTERVENTIONS:
Procedure: Autologous Fat Injection for Rectocele — In this procedure, autologous fat is harvested from the patient's lower abdomen using a multiport cannula. The fat is then processed via centrifugation to separate the viable fat cells, which are emulsified into nanofat. This nanofat is injected into the submucosal layer of the rectocele through the posterior vaginal wall, using an anoscope for guidance. The procedure is intended to reinforce the rectovaginal fascia, alleviate rectocele symptoms such as obstructive defecation and vaginal bulge, and reduce prolapse recurrence.

SUMMARY:
This clinical trial aims to evaluate the effectiveness of autologous fat grafting as a novel treatment for rectocele, a condition characterized by the herniation of rectal tissue into the posterior vaginal wall. Women aged 18 to 60 years with mild to moderate rectocele, presenting with symptoms such as obstructive defecation or vaginal bulge, will undergo submucosal fat injections. The study will assess the procedure's ability to alleviate symptoms and reduce prolapse recurrence. This prospective, single-arm trial will be conducted at Cairo University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 60 years.
* Diagnosis of rectocele confirmed by defecography, with a rectocele size of 2 cm (mild) to 4 cm (moderate).
* Presenting with symptoms of obstructive defecation syndrome, including constipation, incomplete defecation, and/or vaginal bulge.
* Able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients who have previously undergone surgical repair of rectocele.
* Presence of thrombosed hemorrhoids.
* History of sclerotherapy injection for rectocele.
* Diagnosis of anal stenosis.
* History of coagulopathy or current use of anticoagulant or antiplatelet medications.
* Refusal or inability to provide informed consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients ageing from 18 to 60 years presenting to general surgery department of Cairo university hospitals complaining of chronic constipation or obstructed defecation syndrome posterior with posterior vaginal bulge and diagnosed with rectocele
Enrollment: 25 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Reduction in Rectocele Size | 6 months post-procedure
  The outcome will assess the reduction in rectocele size, measured by clinical examination and defecography. Improvement in rectocele grade will be quantified using a standardized rectocele grading scale.
  Rectocele Grading Scale:
  Grade 0: No prolapse of the rectal wall into the vaginal canal. Grade 1: Mild prolapse, where the rectal wall descends slightly into the vaginal canal, typically during straining, but does not reach the vaginal introitus.
  Grade 2: Moderate prolapse, where the rectal wall descends to the level of the vaginal introitus during straining or bowel movements.
  Grade 3: Severe prolapse, where the rectal wall protrudes beyond the vaginal introitus, visible externally, especially during straining.
  This scale would be used to assess the reduction in rectocele size over time as part of your primary outcome. You can adjust the wording in the outcome measure description to reflect this specific scale.
Symptom Relief | 6 months post-procedure
  In this we will evaluate the patient's relief from rectocele-associated symptoms, including vaginal bulge and obstructive defecation. This will be assessed using the Pelvic Floor Distress Inventory-20 (PFDI-20) questionnaire. The PFDI-20 measures the severity of pelvic floor symptoms on a scale of 0 to 4 for each item, with higher scores indicating greater distress.
  Unit of Measure: PFDI-20 Symptom Score (0-100, where 0 represents no distress and 100 represents maximum distress)

SECONDARY OUTCOMES:
Rate of Recurrence of Rectocele | 6 months post-procedure
  This outcome will track the recurrence of rectocele after the autologous fat injection procedure. Recurrence will be defined as the reappearance of rectocele symptoms or the identification of prolapse on clinical examination or defecography.
Postoperative Pain | Up to 1 week post-procedure
  This outcome will assess postoperative pain and discomfort using a standardized pain scale (e.g., Visual Analog Scale) at regular intervals. It will evaluate both the intensity and duration of pain following the fat injection procedure.
  Visual Analog Scale (VAS) for Pain:
  The Visual Analog Scale (VAS) is a tool used to measure pain intensity. It consists of a horizontal line, typically 10 cm in length, with the following markers:
  0 cm: No Pain 5 cm: Moderate Pain 10 cm: Worst Pain Imaginable Participants will be asked to mark a point on the line that best represents their level of pain. The distance from the "No Pain" end to the mark is measured in centimeters to give a quantitative assessment of pain intensity.
  Interpretation:
  0 cm: No Pain 1-3 cm: Mild Pain 4-6 cm: Moderate Pain 7-9 cm: Severe Pain 10 cm: Worst Pain Possible

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications will be shared. This includes data on clinical outcomes, participant demographics, and relevant procedural details. Supporting documents, such as the study protocol and statistical analysis plan, will also be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months after publication of the primary results and will be available for 2 years.
Access Criteria: Access to the de-identified dataset will be granted to researchers who provide a methodologically sound proposal, subject to review and approval by the study team. Proposals should be directed to the principal investigator, and approved proposals will require a data use agreement. Data will be shared via secure data-sharing platforms or repositories.